CLINICAL TRIAL: NCT06742255
Title: Stellate Ganglion Block in Longstanding Facial Nerve Palsy Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Remonda zaki abdelnaeem zaki, Resident at anesthesia, intensive care and pain management, at Assiut University, Assiut University
Other Study IDs: Stellate ganglion facial palsy
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Stellate Ganglion; Facial Palsy; Pain Management
Keywords: Stellate gangliom; Facial palsy
MeSH Terms: conditions — Facial Paralysis; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- stellate ganglion block group
  Interventions: Drug: Stellate Ganglion Block
- medical treatment group

INTERVENTIONS:
Drug: Stellate Ganglion Block — Stellate ganglion block is an injection of local anesthetic at the level of the neck to target the stellate ganglion, a sympathetic ganglion to interrupt abnormal autonomically-mediated pain in patients resistant to medical treatment
  Groups: stellate ganglion block group

SUMMARY:
The goal of the present study is to verify the efficacy of stellate ganglion block (SGB) in the treatment of facial pain

ELIGIBILITY:
Inclusion Criteria:

* facial nerve palsy patients

Exclusion Criteria:

1. light of a recent myocardial infarction.
2. anticoagulant use
3. glucoma
4. lateral nerve palsy
5. emphysema
6. cardiac conduction abnormalities
7. active infection, flu, cold
8. uncontrolled cough
9. Fever
10. Very high blood pressure or if you are on blood thinners.
11. allergic reaction to local anesthetics
12. Primary and secondary coagulopathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: facial nerve palsy patients
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Average motor conduction latency in six muscle of the face | 6 month

SECONDARY OUTCOMES:
Improved muscle tone | 6 months
  facial muscles start to regain their strength improvement of muscle tone.

REFERENCES:
- [Background] Piraccini E, Munakomi S, Chang KV. Stellate Ganglion Blocks. 2023 Aug 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507798/ PMID 29939575
- [Background] Wang D. Image Guidance Technologies for Interventional Pain Procedures: Ultrasound, Fluoroscopy, and CT. Curr Pain Headache Rep. 2018 Jan 26;22(1):6. doi: 10.1007/s11916-018-0660-1. PMID 29374352
- [Background] Kapral S, Krafft P, Gosch M, Fleischmann D, Weinstabl C. Ultrasound imaging for stellate ganglion block: direct visualization of puncture site and local anesthetic spread. A pilot study. Reg Anesth. 1995 Jul-Aug;20(4):323-8. PMID 7577781
- [Background] Abdi S, Zhou Y, Patel N, Saini B, Nelson J. A new and easy technique to block the stellate ganglion. Pain Physician. 2004 Jul;7(3):327-31. PMID 16858470
- [Background] Baig S, Moon JY, Shankar H. Review of Sympathetic Blocks: Anatomy, Sonoanatomy, Evidence, and Techniques. Reg Anesth Pain Med. 2017 May/Jun;42(3):377-391. doi: 10.1097/AAP.0000000000000591. PMID 28272291